CLINICAL TRIAL: NCT04730219
Title: An Open Label, Single-arm, Phase 2 Study of Perioperative Tislelizumab Combined With Nab-Paclitaxel Before Cystectomy or Complete TURBT for Patients With Muscle-invasive Urothelial Bladder Cancer.
Brief Title: Perioperative Tislelizumab Combined With Nab-Paclitaxel for Muscle-invasive Urothelial Bladder Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-01
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Muscle Invasive Bladder Cancer; Urothelial Carcinoma
Keywords: neoadjuvant treatment
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — tislelizumab; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab and Nab Paclitaxel (Experimental): Tislelizumab 200mg IV on day 1 in combination with nab paclitaxel 200mg IV on day 2 every 3 weeks for 3 cycles followed by surgery.
  Interventions: Drug: Tislelizumab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg will be administered on Day 1 every 3 weeks for 3 cycles
  Other Names: BGB-A317
Drug: Nab paclitaxel — Nab paclitaxel 200mg will be administered on Day 2 every 3 weeks for 3 cycles

SUMMARY:
This is a phase II study to determine the safety and efficacy of tislelizumab when given in combination with nab-paclitaxel as perioperative treatment in patients with muscle-invasive bladder cancer (MIBC) prior to cystectomy or complete TURBT. Patients will receive treatment with tislelizumab in combination with nab-paclitaxel every 3 weeks for 3 treatment cycles over 9 weeks followed by standard radical cystectomy or complete TURBT.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Age ≥ 18 years.
4. Suitable and planned for complete transurethral resection of bladder tumor or radical cystectomy
5. Histopathologically confirmed urothelial carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) urothelial cell pattern.
6. Clinical stage T2-T4a N0 M0 disease by CT (or MRI). If the clinical stage is T2-4aN1-3M0, it must be judged by the investigator. If it is judged that radical surgery can still be performed, it can be included in the study.
7. Expected survival time is greater than 12 weeks.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 1 or 2.
9. Agree to provide tissue examination specimens (used to detect PD-L1 expression, tumor mutation burden, etc.)
10. The organ function level must meet the following requirements:

    * Hematological indicators: absolute neutrophil count ≥1.5×10^9/L, platelet count ≥80×10^9/L, hemoglobin ≥6.0 g/dL (can be maintained by symptomatic treatment);
    * Liver function: total bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal value, if there is intrahepatic transaminase ≤ 5 times the upper limit of normal value;
    * Renal function: creatinine ≤ 2 times the upper limit of normal, and creatinine clearance ≥ 30 ml/min;

Exclusion Criteria:

1. Receive live attenuated vaccines within 4 weeks before treatment or plan to receive live attenuated vaccines during the study period.
2. Active, known or suspected autoimmune diseases.
3. Known history of primary immunodeficiency.
4. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
5. Female patients who are pregnant or breastfeeding.
6. Untreated acute or chronic active hepatitis B or C infection. In the case of patients receiving antiviral therapy, the doctor will judge whether they are eligible for enrollment according to the individual conditions of the patient while monitoring the virus copy number.
7. Have used immunosuppressive drugs in the past 4 weeks before starting treatment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (that is, prednisolone or equivalent physiological doses of no more than 10 mg/day) Other corticosteroids).
8. Those who are known or suspected to be allergic to tislelizumab and nab paclitaxel.
9. Have a clear history of active tuberculosis.
10. Have received PD-1/PD-L1/CTLA-4 antibody or other immunotherapy in the past.
11. Those who are participating in other clinical research.
12. Reproductive men or women who are likely to become pregnant have not taken reliable contraceptive measures.
13. Uncontrolled concurrent diseases include but are not limited to:

    * HIV-infected persons (HIV antibody positive).
    * Serious infections that are active or poorly clinically controlled.
    * There are serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [ie refers to After drug treatment, it is still greater than or equal to CTCAE Grade 2 hypertension]) evidence.
    * Active bleeding or new thrombotic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response (cCR) rate | At the time of complete transurethral resection of bladder tumor or radical cystectomy (within 12 weeks of the first dose of tislelizumab)
  defined as the absence of tumor residual confirmed by surgery (RC-PLND or complete TURBT), negative urine cytology and no evidence of lymph nodes or distant metastasis on imaging.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At the time of complete transurethral resection of bladder tumor or radical cystectomy (within 12 weeks of the first dose of tislelizumab)
  defined as the proportion of patients who have a partial or complete response to therapy.
Event-free survival (EFS) | up to 3 years
  defined from D1 of neoadjuvant treatment until progression (in those who progress prior to surgery) or until recurrence (post-surgery) or until death as a result of any cause.
Overall Survival (OS) | up to 3 years
  defined as the number of days from study entry to death. Individuals who are alive at last contact will be censored on the date of last contact.
Disease-specific survival (DSS) | up to 3 years
  DSS was documented from the date of initial treatment till the date of the disease-related death.
Number of adverse events and severity by grade (CTCAE) | up to 1 years
  Safety and toxicity will be characterized according to the reported adverse event (AE) profile using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0, as well as a patient questionnaire derived from the Patient Reported Outcomes (PRO)-CTCAE and Patient Reported Outcomes Measurement Information System (PROMIS).

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Shen C, Chai W, Han J, Zhang Z, Liu X, Yang S, Wang Y, Wang D, Wan F, Fan Z, Hu H. Identification and validation of a dysregulated TME-related gene signature for predicting prognosis, and immunological properties in bladder cancer. Front Immunol. 2023 Oct 27;14:1213947. doi: 10.3389/fimmu.2023.1213947. eCollection 2023. PMID 37965307
- [Derived] Shen C, Bi Y, Chai W, Zhang Z, Yang S, Liu Y, Wu Z, Peng F, Fan Z, Hu H. Construction and validation of a metabolism-associated gene signature for predicting the prognosis, immune landscape, and drug sensitivity in bladder cancer. BMC Med Genomics. 2023 Oct 26;16(1):264. doi: 10.1186/s12920-023-01678-6. PMID 37880682